CLINICAL TRIAL: NCT03684980
Title: LTA Pilot Study of Glucarpidase in Patients With Central Nervous System Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-410
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Central Nervous System Lymphoma
Keywords: Voraxaze (glucarpidase); B-cell non-Hodgkin"s lymphoma involving the brain; B-cell non-Hodgkin"s lymphoma involving spinal cord, and/or leptomeningeal space
MeSH Terms: interventions — Methotrexate; Rituximab; Leucovorin; glucarpidase

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized, pilot study of Voraxaze administered following standard of care MTX and rituximab in patients with CNS lymphoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A - Rituximab + MTX + Glucarpidase (Experimental): Patients will receive rituximab Day 1 (+/- 7 days) and MTX Day 2 (+/- 7 days) as per standard of care. Voraxaze will be administered each cycle 24 hours (+/- 2 h) after start of MTX infusion. Dose of Voraxaze will be 2000 units during cycles 1-4, and 1000 units during cycles 5-8. Patients will be treated with rituximab 500 mg/m^2. (Cohort A) will receive MTX 3 g/m2. Patients will also receive standard of care leucovorin rescue starting at least 24 hours after MTX and 2 hours after Voraxaze. Cycles will be 14 days long.
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: leucovorin; Drug: Glucarpidase
- Arm B - Rituximab + MTX + Glucarpidase (Experimental): Patients will receive up to 8 cycles of treatment consisting of rituximab Day 1 (+/- 7 days) and MTX Day 2 (+/- 7 days) as per standard of care. Voraxaze will be administered each cycle 24 hours (+/- 2 h) after start of MTX infusion. Dose of Voraxaze will be 2000 units during cycles 1-4, and 1000 units during cycles 5-8. Patients will be treated with rituximab 500 mg/m^2. (Cohort B) will receive MTX 8 g/m2. Patients will also receive standard of care leucovorin rescue starting at least 24 hours after MTX and 2 hours after Voraxaze. Cycles will be 14 days long.
  Interventions: Drug: Rituximab; Drug: Glucarpidase
- Arm C - HD-MTX (Arm Outpatient MTX Therapy in times of COVID-19) (Experimental): MTX ≤ 3.5 g/m2 will be administered on Day 1, along with pre- and post- hydration. Patients will return on Day 2 for continued hydration and glucarpidase 2000 units. Glucarpidase rapidly and sustainably reduces serum MTX levels >95% without crossing the blood brain barrier, effectively resulting in systemic MTX clearance. Patients will return for bloodwork on Day 3 to document MTX clearance. Arm Outpatient MTX Therapy in times of COVID-19 will only be a single-institution arm, only open at Memorial Sloan Kettering Cancer Center.
  Interventions: Drug: Methotrexate; Drug: Glucarpidase
- Arm D -Rituximab + MTX + Glucarpidase (Experimental): Up to 12 patients will be included in Arm D of this study. Cycles will be 14 days long. All patients will receive MTX 3.5 g/m2 administered Day 1 of each cycle (+/- 7 days, a minimum of 14 days required between doses). Glucarpidase will be administered 24 hours (+/- 2 hr) after start of MTX infusion except in cycles 1-2 of Cohort B. Dose of glucarpidase will be 2000 units in Cohort A (first 4 patients) and 1000 units in Cohort B (remaining 8 patients). Patients in Arm D will receive 8 cycles of treatment. Cycles 1 and 2 will be administered in patient while Cycles 3-8 may be in the outpatient setting. Concurrent chemotherapy such as vincristine, procarbazine, and/or ibrutinib may be administered at the investigator's discretion and in accordance with standard of care. In Cohort B, all cycles will be administered with rituximab 500 mg/m2. Rituximab should be administered prior to glucarpidase (window -4 days).
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: Glucarpidase
- Arm E-glucarpidase 1000u + MTX (Experimental): Study treatment consists of glucarpidase 1000u, to be administered at least 24 hours after start of standard of care MTX. Patients will have a standard of care methotrexate level drawn within 6 hours of planned glucarpidase administration to confirm eligibility (must reflect MTX > 100 nmol/L)
  Interventions: Drug: Methotrexate; Drug: Glucarpidase

INTERVENTIONS:
Drug: Methotrexate — (Cohort A) will receive MTX 3 g/m2 or (Cohort B) will receive MTX 8 g/m^2 (Cohort E) will receive MTX ≤ 3.5 g/ m2
  Arms: Arm A - Rituximab + MTX + Glucarpidase; Arm C - HD-MTX (Arm Outpatient MTX Therapy in times of COVID-19); Arm D -Rituximab + MTX + Glucarpidase; Arm E-glucarpidase 1000u + MTX
Drug: Rituximab — Patients will be treated with rituximab 500 mg/m^2.
  Arms: Arm A - Rituximab + MTX + Glucarpidase; Arm B - Rituximab + MTX + Glucarpidase; Arm D -Rituximab + MTX + Glucarpidase
Drug: leucovorin — Patients will also receive standard of care leucovorin rescue starting at least 24 hours after MTX and 2 hours after Voraxaze. Cycles will be 14 days long.
  Arms: Arm A - Rituximab + MTX + Glucarpidase
Drug: Glucarpidase — Glucarpidase 2000 units. Arm E 1000 units.
  Other Names: Voraxaze

SUMMARY:
The purpose of this study is to test the effects of a drug called Voraxaze when it's routinely given in combination with methotrexate and rituximab, the standard treatment for CNSL.

ELIGIBILITY:
Inclusion Criteria:

Arm A:

* Histologically documented B-cell non-Hodgkin"s lymphoma involving the brain, spinal cord, and/or leptomeningeal space.

  °Patients in whom the type of lymphoma could not be determined or is unknown (e.g., not enough tissue for further analysis) are assumed to have a B cell lymphoma and are eligible
* Patients with parenchymal lesions must have received no more than two cycles of treatment for treatment of CNS lymphoma or have unequivocal evidence of disease progression on imaging (MRI of the brain/spine or CT head) 28 days prior to study registration. For patients with leptomeningeal disease only, CSF cytology must document lymphoma cells and/or imaging findings must be consistent with CSF disease 28 days prior to study registration (at the discretion of the investigator).
* Patients who have already received two doses of treatment of CNS lymphoma are eligible for enrollment.
* (Arm A only) as long as they are planned for at least 6 additional doses of methotrexate. Patients must not have evidence of systemic non-Hodgkin lymphoma requiring active treatment.
* Men and woman must be at least 18 years of age on the day of consenting to the study.
* Patients must have a Karnofsky Performance Status (KPS) ≥ 50 (See Appendix 2).
* Patients must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests.
* Patients must have adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L;
  * Platelets ≥ 100 x 10^9/L and no platelet transfusion within the past 28 days prior to study registration;
  * Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cells (RBC) transfusion within the past 28 days prior to study registration;
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal;
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal;
  * Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome;
  * CrCl ≥ 60 mL/min using the Cockcroft-Gault equation. Men: CrCl (min/mL) = (140-age) X (actual weight in kg) / 72 X serum creatinine (mg/dL) Women: CrCl (mL/min) = (140-age) X (actual weight in kg) X 0.85 / 72 X serum creatinine (mg/dL)
* Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose.
* Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry.
* Patients must be able to tolerate MRI/CT scans.
* Patients must be able to tolerate lumbar puncture and/or Ommaya taps.
* Participants must have recovered to grade 1 toxicity from prior therapy. NOTE: Patients who have initiated and received up to two cycles of treatment will NOT be excluded from study Arm A as long as all pretreatment assessments have been completed within 28 days of trial initiation.

Arms B and D:

* Histologically documented B-cell non-Hodgkin's lymphoma involving the brain, spinal cord, and/or leptomeningeal space

  ° Patients in whom the type of lymphoma could not be determined or is unknown (e.g., not enough tissue for further analysis) are assumed to have a B cell lymphoma and are eligible
* Patients must be treatment naïve or have unequivocal evidence of disease progression on imaging (MRI of the brain/spine or CT head) 28 days prior to initiation of MTX. For patients with leptomeningeal disease only, CSF cytology must document lymphoma cells and/or imaging findings must be consistent with CSF disease 28 days prior to initiation of MTX. (at the discretion of the investigator)
* Patients must not have evidence of systemic non-Hodgkin lymphoma requiring active treatment
* Men and woman must be at least 18 years of age on the day of consenting to the study
* Patients must have a Karnofsky Performance Status (KPS) >/= 70 or >/= 50 if KPS is due to a neurologic deficit attributed to active disease
* Patients must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests
* Patients must have adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) >/= 1.0 x 10^9/L
  * Platelets >/= 100 x 10^9/L and no platelet transfusion within the past 28 days prior to study registration
  * Hemoglobin (Hgb) >/= 8g/dL and no red blood cells (RBC) transfusion within the past 28 days prior to study registration
  * International Normalized Ratio (INR) </= 1.5 and PTT (aPTT) </= 1.5 times the upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 3 times the upper limit of normal
  * Serum bilirubin </= 1.5 times the upper limit of normal; or total bilirubin </= 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome
  * CrCl >/= 60 mL/min using the Cockcroft-Gault equation Men: CrCl (min/mL) = (140-age) X (actual weight in kg) / 72 X serum creatinine (mg/dL) Women: CrCl (mL/min) = (140-age) X (actual weight in kg) X 0.85 / 72 X serum creatinine (mg/dL)
* Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose.
* Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry
* Patients must be able to tolerate MRI/CT scans
* Patients must be able to tolerate lumbar puncture and/or Ommaya taps
* Participants must have recovered to grade 1 toxicity from prior therapy
* Patients with ocular manifestation of systemic lymphoma are allowed if repeat ophthalmologic exam is planned for the end of therapy. If ocular disease remains present, ocular-directed therapy may be administered after treatment with methotrexate.
* Patients must be able to tolerate po hydration (Arm D only)

NOTE: Prior autologous stem cell transplant as well as prior radiation to the CNS does NOT prevent patients from enrollment into the trial.

Arm Outpatient MTX Therapy in times of COVID-19:

* Patients eligible for inclusion in this arm must be eligible for inpatient MTX administration for treatment of CNS lymphoma. Patients should have received prior MTX therapy without major adverse events.
* Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry.

Arm E:

* Documented history of CNS lymphoma, appropriate for standard of care inpatient MTX administration as determined by their treating physician
* Men and woman must be at least 18 years of age on the day of consenting to the study.
* Patients must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests.
* Patients must meet at least ONE of the following additional criteria

  * MTX >100 nmol/L ≥ 72 hours after initiation of MTX
  * History of prolonged MTX clearance (≥ 72 hours) after prior MTX administration of equal or higher dose (g/m2)
  * CrCl < 60 ml/min calculated by Cockroft-Gault equation oHistory of MTX-related toxicity, CTCAE v5 grade 2 or higher (must have recovered to a grade 1 toxicity)

Exclusion Criteria:

Arms A, B and D:

* Patient with SCNSL requiring treatment for extra-CNS disease are excluded.
* Patient concurrently using other approved or investigational antineoplastic agents.
* Patient has received chemotherapy, monoclonal antibodies or targeted anticancer therapy ≤ 4 weeks or 5 half-lives, whichever is shorter, or 6 weeks for nitrosoureas or mitomycin-C prior to starting the study drug, or the patient has not recovered from the side effects of such therapy. Exceptions are allowed for rituximab and methotrexate for patients enrolling Arm A as long as patients have recovered from side effects.
* Patient has received external beam radiation therapy to the CNS within 28 days of the first dose of the study drug.
* Patient has an active concurrent malignancy requiring active therapy.
* The patient has been treated with radio- or toxin-immunoconjugates within 70 days of the first dose of the study drug.
* Patient weighs <40kg
* Patient is allergic to components of the study drug.
* Patient is known to have human immunodeficiency virus (HIV) infection.
* Patient is known to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests.
* Severe, active medical co-morbidity such as unstable angina and/or congestive heart failure, coronary artery disease, significant abnormalities on electrocardiogram (EKG), uncontrolled or symptomatic arrhythmias or valvular disease; active infection, severe chronic obstructive pulmonary disease or other respiratory illness, hepatic insufficiency, known pre-existing immunodeficiency as seen in organ transplant recipients, renal failure with CrCl <60 mL/min.
* Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject"s safety or put the study outcomes at undue risk.
* Patient has large pleural or ascetic fluid collection.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Prior severe allergic reaction to any of the study drugs that cannot be resolved with medication.
* Patient has undergone prior allogenic stem cell transplant (autologous stem cell transplant is NOT an exclusion).

Arm Outpatient MTX Therapy in times of COVID-19:

Patients eligible for this arm must not meet any of the following criteria:

* Patients with SCNSL requiring treatment for extra-CNS disease are excluded.
* Patients weighing <40kg
* Inadequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) </= 0.5 x 10^9/L
  * Platelets </= 75 x 10^9/L
  * Hemoglobin (Hgb) </= 8 g/dL
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >/= 3 times the upper limit of normal
  * Serum bilirubin >/= 1.5 times the upper limit of normal; or total bilirubin >/= 3 times the upper limit of normal with direct bilirubin outside of the normal range in patients with well documented Gilbert Syndrome
  * Creatinine >/= 1.3 mg/dL
* Patients allergic to components of the study drug.
* Patients with severe, active medical co-morbidity such as unstable angina and/or congestive heart failure, coronary artery disease, significant abnormalities on electrocardiogram (EKG), uncontrolled or symptomatic arrhythmias or valvular disease; active infection, severe chronic obstructive pulmonary disease or other respiratory illness, hepatic insufficiency, known pre-existing immunodeficiency as seen in organ transplant recipients, renal failure with creatinine >/= 1.3 mg/dL.
* Patients with a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk
* Patients with large pleural or ascetic fluid collection
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic. Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose

Arm E:

Patients eligible for this arm must not meet any of the following criteria:

* Weight <40kg
* Prior severe allergic reaction to methotrexate or glucarpidase that cannot be resolved withmedication.
* Severe, active medical co-morbidity such as unstable angina and/or congestive heart failure, coronary artery disease, significant abnormalities on electrocardiogram (EKG), uncontrolled or symptomatic arrhythmias or valvular disease; active uncontrolled infection, severe chronic obstructive pulmonary disease or other respiratory illness, hepatic insufficiency
* Patient has a life-threatening illness, medical condition, or organ system dysfunctionthat, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk.
* Presence of large pleural or ascetic fluid collection.
* Treatment with MTX dose greater than 8 g/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
number of patients that have significant reduction of serum methotrexate levels | 1 year
  All serum samples will be tested via MTX immunoassay (measures MTX levels in addition to byproducts) as well as HPLC or mass spectroscopy which will reveal plasma concentrations of MTX and DAMPA separately.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Schaff, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dana Farber Cancer Institute (Data Collection and Specimen Analysis), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic (Data Collection and Specimen Collection), Cleveland, Ohio

REFERENCES:
- [Derived] Schaff LR, Carlow D, Schofield R, Wongchai V, Madzsar J, Hyde A, Reiner AS, Panageas KS, DeAngelis LM, Mellinghoff IK, Lobbous M, Nabors LB, Grommes C. Low-Dose Planned Glucarpidase Allows Safe Outpatient High-Dose Methotrexate Treatment for CNS Lymphoma. JCO Oncol Pract. 2024 Oct;20(10):1384-1390. doi: 10.1200/OP.24.00080. Epub 2024 Jun 25. PMID 38917404
- [Derived] Schaff LR, Lobbous M, Carlow D, Schofield R, Gavrilovic IT, Miller AM, Stone JB, Piotrowski AF, Sener U, Skakodub A, Acosta EP, Ryan KJ, Mellinghoff IK, DeAngelis LM, Nabors LB, Grommes C. Routine use of low-dose glucarpidase following high-dose methotrexate in adult patients with CNS lymphoma: an open-label, multi-center phase I study. BMC Cancer. 2022 Jan 13;22(1):60. doi: 10.1186/s12885-021-09164-x. PMID 35027038
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm